CLINICAL TRIAL: NCT05630313
Title: Gene Sequencing as a Strategy for Identifying Genetic Factors Associated With Serious Adverse Events After Covid-19 Vaccines in Use in Brazil
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 001/2022
Record Dates: First submitted 2022-11-23; First posted 2022-11-29 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Vaccine-induced Thrombotic Thrombocytopenia Syndrome; Guillain-Barre Syndrome; Acute Disseminated Encephalomyelitis; Transverse Myelitis
Keywords: Vaccine-induced thrombotic thrombocytopenia; Guillain-Barre Syndrome; Acute Disseminated Encephalomyelitis; Transverse Myelitis; Covid-19 vaccine; Seriuos Adverse Events
MeSH Terms: conditions — Guillain-Barre Syndrome; Encephalomyelitis, Acute Disseminated; Myelitis, Transverse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol proposes to investigate genetic factors that may be involved in the pathogenesis of adverse events of interest with selected covid-19 vaccines: vaccine-induced immune thrombotic thrombocytopenia, and neurological adverse events, such as Guillain-Barré syndrome, acute disseminated encephalomyelitis and transverse myelitis, with the intention of identifying useful biomarkers in identifying people at higher risk, thus reducing the occurrence of these serious adverse events (SAE).

DETAILED DESCRIPTION:
Participants higher than 5 years old with no maximum age limit and both sexes, who had a serious adverse event after vaccination against Covid-19, such as Guillain-Barré syndrome, vaccine-induced immune thrombotic thrombocytopenia, transverse myelitis and Acute disseminated encephalomyelitis. Parents, siblings and/or sons of cases with SAE will have biological samples collected and stored; depending on the result of the study, they may have their samples analyzed later.

ELIGIBILITY:
Inclusion Criteria:

* Sign the ICF by the subject or the subject's legally acceptable representative;
* Sign the ICF by the participant's family member;
* Proven vaccination with one of the vaccines for COVID-19 available by the PNI, containing information on the date of application, type (manufacturer) of vaccine received and batch (desirable);
* Meet the minimum criteria for a level of certainty 3, 2 or 1 in Brighton Collaboration for vaccine-induced immune thrombotic thrombocytopenia as described in 3.2.1.1 OR,
* Meet the minimum criteria for a level of certainty 3, 2 or 1 in Brighton Collaboration for Guillain-Barré syndrome as described in 3.2.1.3 OR,
* Meet the minimum criteria for a level of certainty 3, 2 or 1 in Brighton Collaboration for Acute Disseminated Encephalomyelitis as described in 3.2.1.4 OR,
* Meet the minimum criteria for a level of certainty 3, 2 or 1 in Brighton Collaboration for Transverse Myelitis as described in 3.2.1.5 OR,
* Be classified in the causality categories adopted by the PNI/MS, namely: A1, B1 or B2.

Exclusion Criteria:

* Reports in which it is not possible to retrieve the clinical/laboratory data necessary for evaluation, due to inadequate filling of the notification or unavailability of data;
* Cases of death in which there are no samples available and/or suitable for carrying out the analyzes defined in the protocol;
* Cases in which another diagnosis is made for the adverse event of interest, being discarded as a SAE;
* Cases classified in causality categories (PNI/MS) as A2, A3, A4, C or D;
* Refusal to sign the informed consent form;

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects more than 5 years to no limit maximum age, both sex, which have presented the protocol interest SAE (vaccine-induced immune thrombotic thrombocytopenia, Guillain-Barré syndrome, Acute Disseminated Encephalomyelitis, Transverse Myelitis) can be arrolled. First-degree relatives, primarily parents and/or siblings, will have biological samples collected and stored to be used for future genomic sequencing, if genetic alterations are identified in their relatives who had SAE.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Genomic evaluation | March, 2023.
  Identify if any genetic marker is envolved in the serious adverse event pathogenesis induced by covid-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia de Oliveira, MD, Principal Investigator — Instituto Fernandes Figueira
Locations (1):
- Unidade de Ensaios Clínicos para Imunobiológicos (UECI), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No